CLINICAL TRIAL: NCT05457816
Title: Genetic and Social Network Correlates of Rheumatoid Arthritis Outcomes in Hispanic Populations: A Prospective Study
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000912; 000912-HG
Record Dates: First submitted 2022-07-09; First posted 2022-07-14 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Joint; Pain; Health Service Use; Immigrants; Natural History
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- family members: family members of those with rheumatoid arthritis
- rheumatoid arthritis: persons with rheumatoid arthritis

SUMMARY:
Background:

Rheumatoid arthritis (RA) is more severe in Hispanic people. Genetics plays a role. But social issues may also lead to more severe RA in Hispanics. Some Hispanics may not seek help for early symptoms. Support from family and friends may persuade people to seek treatment earlier. Researchers want to learn more about how social factors affect RA in Hispanics.

Objective:

This natural history study will explore genetic and social factors related to RA in Hispanic families.

Eligibility: People aged 18 years or older of Hispanic/Latino heritage. They may have RA or RA symptoms; they may also have a relative or partner with RA or RA symptoms.

Design:

Participants will receive an email or text with a link to a 30-minute online survey. They will answer questions about these things:

Physical and emotional health

How health problems affect their life

Family history of RA and other conditions

Cultural identity and language preference

Participants may also answer these questions in a phone call or an in-person interview.

Participants will be asked to list people in their social network. They will answer questions about those relationships. They will be asked if they want to invite their family and friends to participate in the study.

If more than 1 person from a participant s family takes part in the study, they may be invited for an interview. They will answer questions about how arthritis pain affects their mind and body.

Participants will give a sample of saliva. They will spit into a vial. They will mail it in using a prepaid label.

DETAILED DESCRIPTION:
Study Description:

Adult participants of Hispanic origin experiencing rheumatoid arthritis (RA) symptoms and their family members will be invited to participate in surveys and interviews to assess RA severity (affected individuals only), functional limitations, psychological well-being, use of health service, and family networks. Genotyping will be performed on saliva samples collected from consenting participants to evaluate genetic risk of severe RA in the population under study.

Objectives:

The primary objective is to identify the interpersonal mechanisms underlying RA-related health communication and health service use in Hispanic populations. The secondary objective is to characterize genetic risk of severe RA in Hispanic populations and determine how interpersonal mechanisms moderate such genetic risk.

Endpoints:

Primary Endpoint: Evaluate the associations between structural properties of the participants personal networks and RA-related health communication and use of health service

Secondary Endpoint: Evaluate the associations between family networks, RA-related health communication and use of health service, and RA severity across levels of genetic susceptibility

ELIGIBILITY:
* INCLUSION CRITERIA:

Consistent with the study objective, to be eligible to participate in this study, an individual must meet all of the following:

* Age 18 and over;
* Able to speak either English or Spanish;
* Of Hispanic/Latino heritage (regardless of country of origin);
* Meeting one of the following: (a) has RA or RA symptoms, (b) has at least one biological kin who has RA or RA symptoms, (c) has a spouse/partner who has RA or RA symptoms. It is not required to have an official diagnosis or records of symptoms. The screening questionnaire will screen prospective participants for either a confirmed diagnosis of RA or presence of inflammatory polyarthritis (pain, swelling and stiffness in three or more joints), which is the evaluation criterion for suspected RA in absence of laboratory testing, for themselves or their biological relatives or spouse/partner;
* Able and willing to give written informed consent.

EXCLUSION CRITERIA:

This is a study being conducted at NHGRI s intramural research program. Therefore, NHGRI staff will be excluded from as a safeguard against the risk of ethical concerns.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants of Hispanic origin experiencing rheumatoid arthritis (RA) symptoms and their family members
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Family networks | One time
  Evaluate the associations between family networks, RA-related health communication and use of health service, and RA severity across levels of genetic susceptibility

CONTACTS AND LOCATIONS:
Overall Officials: Jielu Lin, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (2):
- United States (2):
  - National Human Genome Research Institute (NHGRI), Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000912-HG.html